CLINICAL TRIAL: NCT06391879
Title: Establishment of a Multidimensional Prediction Model for the Natural Course of VHL Disease-related Renal Cell Carcinoma Based on Accurate Genotyping: a Population-based Study
Brief Title: Establishment of a Multidimensional Prediction Model for the Natural Course of VHL Disease-related Renal Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, GONG Kan, Chief physician, Peking University First Hospital
Other Study IDs: 2023#395-002
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: VHL Syndrome; Renal Cell Carcinoma
Keywords: VHL; VHL syndrome; Renal cell carcinoma
MeSH Terms: conditions — von Hippel-Lindau Disease; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VHL-related RCC cohort: This cohort incorporates subjects with VHL-related renal cell carcinoma.
  Interventions: Genetic: Single cell sequencing, whole genome and metabolomic sequencing

INTERVENTIONS:
Genetic: Single cell sequencing, whole genome and metabolomic sequencing — The blood specimen of subjects in this cohort would be collected to conduct single cell sequencing, whole genome and metabolomic sequencing.

SUMMARY:
VHL syndrome is a rare hereditary tumor syndrome caused by mutation of tumor suppressor gene VHL. One of the most important clinical manifestations and main cause of death is VHL-related renal cell carcinoma (RCC). Facing the challenges of multilesion of both kidneys, slow progress and life-long repeated surgeries in VHL-related RCC, individualized prediction of the best surgical treatment time and reduction of times of surgeries are very important to improve the prognosis of patients with VHL syndrome. Therefore, there is an urgent need to establish a more effective and accurate prediction model for the natural course of VHL syndrome. This cohort-study aims to retrospectively and prospectively analyze the factors related to the natural course of VHL-related RCC. At the same time, some patients were selected for prospectively continuous molecular evolution dynamic monitoring after comprehensively considering the results of single cell sequencing, whole genome and metabonomic sequencing. This study will provide scientific basis for accurate diagnosis and treatment of natural course of VHL-related RCC.

DETAILED DESCRIPTION:
VHL syndrome is a rare hereditary tumor syndrome caused by mutation of tumor suppressor gene VHL. One of the most important clinical manifestations and main cause of death is VHL-related renal cell carcinoma (RCC). Previous small sample studies have confirmed that the natural course of VHL-related RCC is different from that of sporadic RCC. Facing the challenges of multilesion of both kidneys, slow progress and life-long repeated surgeries in VHL-related RCC, individualized prediction of the best surgical treatment time and reduction of times of surgeries are very important to improve the prognosis of patients with VHL-related RCC. Therefore, there is an urgent need to establish a more effective and accurate prediction model for the natural course of VHL syndrome. Based on the previous establishment of the largest biobank of VHL syndrome in Asia, as well as the unique characteristics and genotype-phenotypic relationship of patients in Chinese population, this cohort-study aims to retrospectively and prospectively analyze the factors related to the natural course of VHL-related RCC. At the same time, some patients were selected for prospectively continuous molecular evolution dynamic monitoring after comprehensively considering the results of single cell sequencing, whole genome and metabonomic sequencing. This study will systematically analyze the specific molecular characteristic and evolution of VHL-related different from sporadic RCC, reveal new specific driving genes and their molecular regulatory mechanisms, and establish a multi-dimensional prediction model of natural course of VHL-related RCC based on accurate genotyping. It will provide scientific basis for accurate diagnosis and treatment of natural course of VHL-related RCC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of VHL syndrome based on clinical diagnostic criteria or genetic test results of syndrome
* Upon enrollment, multiple organ assessments for VHL syndrome should be completed, including fundus examination, CT/MR examination of the brain, spinal cord, and abdominal and pelvic organs.
* If subjects have undergone surgery for renal tumors, the follow-up observation time in each branch center before surgery should be more than 12 months, and imaging examinations should be performed at least once every 6 months.

Exclusion Criteria:

* Do not meet the clinical diagnostic criteria for VHL disease or the genetic test is negative
* Other hereditary RCC syndromes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the previous establishment of the largest biobank of VHL syndrome in Asia, as well as the unique characteristics and genotype-phenotypic relationship of patients in Chinese population, this cohort-study aims to retrospectively and prospectively incorporated patients with VHL-related RCC.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Tumor growth rate | From date of diagnosis of the VHL-related RCC until the date of surgical treatment, death from any cause or the date of last follow-up, whichever came first, assessed up to 60 years.
  The tumor size was measured annually and the tumor growth rate was calculated.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of diagnosis of the VHL-related RCC until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 20 years.
  OS was calculated as the time interval from the diagnosis of the VHL-related RCC to death or the time to the last follow-up.
Cancer-specific survival (CSS) | From date of diagnosis of the VHL-related RCC until the date of death from the same disease or the date of last follow-up, whichever came first, assessed up to 20 years.
  CSS was calculated as the time interval from the diagnosis of the VHL-related RCC to death from the same disease or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kan Gong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China